CLINICAL TRIAL: NCT01448993
Title: Effect Of Azithromycin On Oesophageal Function In Patients With Dysphagia Or Gastro-Oesophageal Reflux Associated With Frequent Oesophageal Hypomotility
Brief Title: Effect of Azithromycin on Oesophageal Hypomotility
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JAFAR JAFARI (Other)
Responsible Party: Sponsor-Investigator, JAFAR JAFARI, CLINICAL RESEARCH FELLOW, Queen Mary University of London
Organization: Queen Mary University of London (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BICMS/PR/11/127
Record Dates: First submitted 2011-09-30; First posted 2011-10-07 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Esophageal Motility Disorders
MeSH Terms: conditions — Esophageal Motility Disorders | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Taking placebo 3 times per week for four weeks
  Interventions: Drug: Placebo
- AZI (Active Comparator)
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Taking 250mg azithromycin 3 times per week in alternate days.
  Arms: AZI
Drug: Placebo
  Arms: Placebo

SUMMARY:
Patients with difficulty in swallowing (dysphagia) or with reflux disease are frequently found to suffer from oesophageal hypomotility (weak contractions).

Oesophageal motility is currently measured using high-resolution manometry (HRM). This technique has a 36 pressure sensors on a plastic tube to record the pressure in side the oesophagus.

Several pharmaceutical agents (prokinetics) can stimulate oesophageal motility. However, use of prokinetics in patients with oesophageal hypomotility led to disappointing results. An explanation for these disappointing results is that inappropriate patients were targeted. The appropriate patient would be the one who still have some viable muscle in the oesophagus that can respond to pharmacological stimuli.

In the process of developing treatment strategies in patients with oesophageal hypomotility, testing the preserved capacity of oesophageal muscles could be useful to predict the response of these patients to prokinetic drugs. The following tests have the potential to reveal the preserved capacity of the oesophageal muscle to respond to stronger/medicinal stimuli.

1. - Multiple rapid swallowing (MRS) of 5ml water boluses stimulates oesophagus. A normal response to MRS requires on the one hand integrity of neural mechanisms and on the other hand a functional oesophageal muscle.
2. - External abdominal compression can increase the resistance to bolus transport via oesophagus. The normal oesophagus produces contractions of higher amplitude and duration in order to maintain a normal bolus transit.
3. - Swallowing bread boluses require stronger oesophageal contractions for a successful bolus transit.

The purpose of the proposed project is to firstly assess the effect of Azithromycin on oesophageal hypomotility and secondly to evaluate the predictive values of the stimulation techniques in predicting the likelihood the positive response to drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects:

   1. Written ICF signed voluntarily before the first trial-related activity.
   2. Subjects male and female within age range of 18-70 years old (extremes included)
   3. BMI <35
2. Patients group:

   1. Written ICF signed voluntarily before the first trial-related activity.
   2. Patients male and female, aged 18-70
   3. Been diagnosed with severe oesophageal hypomotility based on Chicago classification 2011
   4. Must have moderate or severe reflux symptoms and/ or dysphagia, with at least one of these symptoms of moderate severity or worse, and at a minimum average frequency of three days a week during the two weeks prior to the study date
   5. If the subject is a woman of childbearing potential, she

      1. must have a negative urine pregnancy test before the start of treatment (minimum β-Human Chorionic Gonadotropin [HCG] sensitivity of 25 mIU/ml), and
      2. must agree to either use an effective form of birth control (i.e., stabilized on oral contraceptives for at least 1 month or using implanted, transdermal or injected contraceptive hormones, an intra-uterine device, or continuous abstinence from heterosexual sexual contact), or a combination of a barrier method and a spermicidal agent (i.e., cervical cap and spermicidal agent, condom and spermicidal agent, or diaphragm and spermicidal agent),

Exclusion Criteria:

* Healthy subjects:

  1. Any incidental abnormal oesophageal motility finding
  2. History of gastrointestinal symptoms, gastrointestinal tract surgery or other recent abdominal operation within last 3 months.
  3. Major psychiatric, neurological, respiratory, liver, haemorrhagic and cardiac disorders, malignancies
  4. Pregnancy and no wheat allergy
* Patients:

  1. Subjects with a documented history of long segment (>3 cm) Barrett's oesophagus.
  2. Subjects with documented or suspected large (> 3 cm) hiatus hernia.
  3. Subjects with fundoplication, endoscopic anti-reflux procedure or major prior GI surgery.
  4. Subjects with structural abnormalities of oesophagus (ie. Rings and webs, scleroderma)
  5. Severe oesophageal motility disorders other than oesophageal hypomotility (e.g., achalasia, nutcracker oesophagus).
  6. Subjects who suffer from frequent vomiting (>1/week)
  7. Current diagnosis of co-existing psychiatric disease (including alcohol or drug abuse); controlled depression and anxiety are allowed, when treated with at most
  8. Allergy to prokinetic medicine (AZI), gluten or egg, allergy to latex (reflux monitoring catheter has cross reaction with latex)
  9. Patients with concomitant prohibited medications, unless willing or able to withdraw from these medications
  10. Use of prohibited co-medication less than 7 days before the start of the study
  11. Any condition that, in the opinion of the Investigator, would complicate or compromise the trial (e.g., human immunodeficiency virus [HIV] infection, gastroduodenal ulcer) or the well-being of the subject, or evidence of any clinically relevant pathology that could interfere with trial results or put subject safety at risk.
  12. Participation in an investigational drug trial in 30 days prior to enrolment.
  13. Pregnant or breast-feeding subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Effect of Azithromycin on oesophageal peristalstic contraction amplitude in patients with hypomotility | 4 weeks
  The amplitude of peristaltic contractions and also Distal Contractal Integral which summarises the vigour of peristalsis will be measured before and after treatment with Azithromycin. Measurement is performed by oesophageal high resolution manometry. The measures will be compared to decide on the effect oo Azithromycin on oesophageal motility.

SECONDARY OUTCOMES:
Manometric oesophageal body response (amplitude of peristaltic contractions in mmHg and also Distal Contractal Integral in mmHg.cm.second) to solid bolus swallows, MRS and outlet obstruction in healthy subjects and patients with oesophageal hypomotility. | 4 weeks
  The above parameters will be measured before and after treatment with Azithromycin. Measurement is performed by oesophageal high resolution manometry. The measures will be compared to decide on the effect oo Azithromycin on oesophageal motility.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital, London, London, United Kingdom